CLINICAL TRIAL: NCT01118403
Title: Antibiotic Prophylaxis for Early Ventilator-associated Pneumonia in Neurological Patients: A Randomized Trial
Brief Title: Antibiotic Prophylaxis for Early Ventilator-associated Pneumonia in Neurological Patients
Acronym: NAVPRO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: He could not be started due to lack of funds
Sponsor: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 58222
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated pneumonia; Coma; Brain Injuries; Intensive care units; antibiotic prophylaxis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Coma; Brain Injuries | interventions — sultamicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sultamicillin, Antibiotic Prophylaxis (Experimental): Sultamicillin, Antibiotic Prophylaxis
  Interventions: Drug: Sultamicillin
- Placebo (Placebo Comparator): Physiologic Sodium Chloride Solution
  Interventions: Drug: Sultamicillin

INTERVENTIONS:
Drug: Sultamicillin — Ampoules per 1.5 grams, three grams intravenously every 6 hours for 4 doses diluted in physiologic Sodium Chloride Solution
  Other Names: Sulbactam Ampicillin; Unasyn

SUMMARY:
This study seeks to assess whether coma patients really benefit from the use of antibiotics as a prophylactic for reducing the incidence of early ventilator-associated pneumonia in this population group. For this we consider the use of ampicillin sulbactam antibiotic which has a low ability to induce resistance, efficacy and safety observed during the time that has been used, even in patients with neurosurgical pathology, and to be broadly available in our environment.

Our hypothesis is that neurological patients in coma state, requiring mechanical ventilation, the application of antibiotic prophylaxis compared with placebo reduces the incidence of early ventilator-associated pneumonia.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the most common nosocomial infections occur in intensive care units, with frequencies ranging between 15% and 45%, which determine an attributable mortality of 25% to 27%

Patients with compromised state of consciousness brought to mechanical ventilation, have a much higher reported incidence that patients without neurological involvement, reaches between 44 and 70%.

These data have led to plan the implementation of strategies to reduce the incidence of early pneumonia in this population group, to thereby favorably influence the high rates of mortality, morbidity and costs that arise.

Then we design this study to assess whether these patients really benefit from the use of antibiotics as a prophylactic, considering also the high impact that this would have given the high incidence of early ventilator-associated pneumonia in this population group.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to intensive care units,with score in the Glasgow Coma scale less than nine.
* Requiring mechanical ventilation for more than 48 hours
* Includes all patients with structural or metabolic coma

Exclusion Criteria:

* Pregnant women
* History of allergic reactions to ampicillin sulbactam
* Patients admitted as potential organ donors
* Patients with an indication of antibiotic therapy, or who have received more than 2 doses of any antibiotic previously.
* Hospital stay for more than 48 hours before intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Impact of prophylaxis with ampicillin sulbactam versus placebo on the incidence of early ventilator-associated pneumonia | 2 years
  To determine the impact of prophylaxis with ampicillin sulbactam versus placebo on the incidence of early ventilator-associated pneumonia in patients with altered level of consciousness with a score on the Glasgow Coma Scale less than or equal to 8 and requiring mechanical ventilation for more than 48 hours

SECONDARY OUTCOMES:
Effect of antibiotic prophylaxis versus placebo on the incidence of other infections | 2 years
  Compare the effect of antibiotic prophylaxis versus placebo on the incidence of later ventilator-associated pneumonia, as well as in other non-pulmonary infections (catheter sepsis, bacteremia, meningitis, urinary tract infection).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Cadavid, MD, Principal Investigator — Hospital Pablo Tobón Uribe
Locations (1):
- Hospital Pablo Tobón Uribe, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No